CLINICAL TRIAL: NCT06378437
Title: A Phase 1, Open-label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, Pharmacodynamics and Preliminary Efficacy of GLB-001 in Patients With Myeloid Malignancies
Brief Title: A Study of GLB-001 in Patients With Myeloid Malignancies
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hangzhou GluBio Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: GLB-001-02
Record Dates: First submitted 2024-04-18; First posted 2024-04-22 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-03

CONDITIONS: Polycythemia Vera; Essential Thrombocythemia; Myelofibrosis; Myelodysplastic Syndromes; Acute Myeloid Leukemia; Myeloid Malignancy
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential; Primary Myelofibrosis; Myelodysplastic Syndromes; Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Dose Escalation of GLB-001 in Study Participants with PV and ET-Phase 1a (Experimental): Phase 1a (Dose Escalation) will evaluate the safety and tolerability of GLB-001 in PV and ET study participants. A standard 3+3 dose-escalation design will be applied to evaluate a set of dose levels to determine and the maximum tolerated dose (MTD) and/or recommended expansion doses (RED) in PV and ET study participants who are eligible for dose limiting toxicity (DLT) evaluation.
  Interventions: Drug: GLB-001
- Dose Exploration of GLB-001 in Study Participants with MF, LR-MDS, AML and HR-MDS-Phase 1b (Experimental): Phase Ib 1b (Dose Exploration) will utilize a standard 3+3 dose-escalation design to evaluate the safety and tolerability of GLB-001 in MF, LR-MDS, HR-MDS and AML study participants. The starting dose will be selected within the range of tolerated dose levels determined in Phase 1a (Dose escalation).
  Interventions: Drug: GLB-001
- Dose Expansion of GLB-001 in Study Participants with PV, ET, MF, LR-MDS, AML and HR-MDS-Phase 1c (Experimental): Phase 1c (Dose Expansion) will be conducted to further determine the tolerability, efficacy and the recommended phase 2 dose (RP2D) of GLB-001 in study participants with relapsed or refractory or intolerant myeloid malignancies including PV, ET, MF, LR-MDS, HR-MDS and AML.
  Interventions: Drug: GLB-001

INTERVENTIONS:
Drug: GLB-001 — Administered orally according to the assigned treatment schedule
  Other Names: GLB-C183-A-2

SUMMARY:
Study GLB-001-02 is a phase 1, open-label clinical study to evaluate the safety, tolerability, pharmacokinetics (PK), pharmacodynamics (PD) and preliminary efficacy of GLB-001 in study participants with relapsed or refractory or intolerant myeloid malignancies including polycythemia vera (PV), essential thrombocythemia (ET), myelofibrosis (MF), lower-risk myelodysplastic syndrome (LR-MDS), higher-risk myelodysplastic syndromes (HR-MDS), and acute myeloid leukemia (AML). This study consists of 3 parts, dose escalation (Phase 1a), dose exploration (Phase 1b) and dose expansion (Phase 1c). Dose escalation (Phase 1a) and dose exploration (Phase 1b) will evaluate the safety, tolerability, PK, PD and preliminary efficacy of GLB-001, administered orally, in study participants with PV/ET, or study participants with MF/LR-MDS/HR-MDS/AML, respectively. Dose expansion (Phase 1c) will be followed to determine the relationships among dose, exposure, toxicity, tolerability and clinical activity, to identify minimally active dose, and to select the recommended dose(s) for phase 2 study. Approximately 108 study participants may be enrolled in the study.

ELIGIBILITY:
Inclusion Criteria:

* Study participants must understand and voluntarily sign a written informed consent form (ICF) prior to any study-related assessments/procedures being performed.
* Study participants is ≥18 years of age at the time of signing the ICF.
* Study participants with confirmed diagnosis of relapsed or refractory or intolerant myeloid malignancies including PV, ET, primary myelofibrosis (PMF), MDS and AML according to 2022 World Health Organization (WHO) criteria classification, and post-polycythemia vera myelofibrosis (post-PV MF) and post-essential thrombocythemia myelofibrosis (post-ET MF) according to the 2013 IWG-MRT criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0,1 or 2.
* Life expectancy > 3 months.
* Good performance of major organs, including hematology, liver and kidney function, and coagulation. etc.
* Study participants are willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

* Study participants with acute promyelocytic leukemia (APL).
* Receipt of following anticancer medications/therapies prior to the first dose of GLB-001: (1) study participants with PV or ET who received treatment with hydroxyurea within 2 days prior to the first dose, or any other treatment for PV or ET within 7 days prior to first dose of GLB-001, (2) study participants with MF who received any type of treatment for MF within 14 days prior to the first dose, such as chemotherapy, immunotherapy, radiotherapy and erythropoietin, androgens, thrombopoietin or granulocyte colony-stimulating factor, (3) study participants with LR-MDS who received any type of treatment for MDS within 14 days prior to the first dose, (4) study participants with HR-MDS or AML who received chimeric antigen receptor T cell therapy (CAR-T) or other biologic therapy within 28 days prior to the first dose of GLB-001, or received any other anticancer therapies within 14 days prior to the first dose of GLB-001.
* Receipt of any other investigational drug study within 28 days or 5 half-lives of that study drug before the first dose of GLB-001.
* Study participants with unresolved clinically significant non-hematologic toxicities that were ≥ Grade 1 or failed to recover to baseline levels following prior anticancer therapies (with the exception of alopecia or skin hyperpigmentation).
* Study participants who are scheduled to receive other anticancer therapies or other investigational drugs during the study period.
* Study participants with active acute or chronic graft versus host disease (GVHD) requiring systemic immunosuppressive therapy.
* Receipt of autologous stem cell transplantation (ASCT) within the last 3 months prior to the first dose of GLB-001, or allogeneic hematopoietic stem cell transplantation (allo-HSCT) within the last 6 months prior to the first dose of GLB-001.
* Study participants with known active involvement in central nervous system (CNS).
* Study participants with peripheral neuropathy ≥ Grade 2 (Graded according to CTCAE version 5.0).
* Study participants have a history of known malignancy other than the inclusion diagnosis for the past 5 years, with the exception of curatively resected cancer in situ, including cervical carcinoma in situ, basal cell carcinoma of the skin, or prostate cancer in situ, etc.
* QT interval interval > 450 milliseconds (ms) using electrocardiographic (ECG) at screening.
* Study participants have impaired cardiac function or clinically significant cardiac disease at current or within last 6 months.
* Study participants with known active infection of hepatitis B virus (HBV) or hepatitis C virus C (HCV).
* Study participants with known human immunodeficiency virus (HIV) infection.
* Study participants with known life-threatening or clinical significant uncontrolled active systemic infections unrelated to malignant hematologic diseases.
* Study participants with a state condition that may alter affects the absorption, distribution, metabolism and excretion of GLB-001 after judgment of the investigator.
* Medications or supplements that are known to be strong and moderate inhibitors or inducers of cytochrome P-450 isozyme 3A (CYP3A) and/or P-glycoprotein (P-gp), or strong inhibitors or inducers of CYP450 isozyme 2C8 (CYP2C8) within 7 days or 5 half-lives prior to the first dose of GLB-001, whichever is shorter prior to the first dose of GLB-001.
* Study participants who have undergone major surgery within 28 days prior to the first dose of the GLB-001, or unability to recover from effects of surgery.
* Pregnant or lactating women.
* Study participants who have cognitive impairment due to any psychiatric or neurological condition, including epilepsy and dementia, may limit their understanding, performance, and study compliance with the ICF.
* Study participants, in the opinion of the Investigator, who are unsuitable to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2024-05-24 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose-limiting Toxicity (DLT) | Up to 28 days after first dose of study treatment in Phase 1a and Phase 1b
  DLT is defined as the treatment emergent adverse events (TEAEs) meeting protocol specified DLT criteria and occurring within the DLT assessment period.
Maximum Tolerated Dose (MTD) | Up to 1 year in Phase 1a and Phase 1b
  MTD is defined as the highest dose level at which no more than 1 of 6 DLT-evaluable study participants experienced a DLT.
Recommended Expansion Doses (RED) | Up to 1 year in Phase 1a and Phase 1b
  RED will be determined by the safety review committee (SRC) according to the safety, tolerability, PK, PD, and preliminary efficacy of GLB-001 in dose escalation phase and dose exploration phase.
Incidence, Relatedness, Seriousness and Severity of Adverse Events (AEs) | Up to 3 years in Phase 1a and Phase 1b
  AE is any untoward medical occurrence in a study participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment. AE will be graded according to the National Cancer Institute Common Terminology Criteria for AE (NCI CTCAE) version 5.0.
Recommended Phase 2 Dose (RP2D) | Up to 1 year in Phase 1c
  RP2D based on the totality of data across dosing cohorts in the dose escalation, dose exploration and dose expansion phases of the study including PK, PD, safety and efficacy outcomes.
Response Assessment in Study Participants With PV | Up to 3 year in Phase 1c
  Response will be evaluated according to the European Leukemia Net (ELN) and 2013 International Working Group for Myelofibrosis Research and Treatment (IWG-MRT) criteria, including overall response rate (ORR), duration of remission or response (DOR), time to response (TTR), progression-free survival (PFS), percentage of study participants who achieved complete hematologic response (CHR), duration of CHR, percentage of study participants with hematocrit (HCT) <45%, percentage of study participants with >50% change in Myeloproliferative Neoplasm Symptom Assessment Total Symptom Score (MPN-SAF TSS), percentage of study participants who achieve spleen volume reduction of greater than or equal to 35% (SVR35) from baseline, duration of SVR35 (DoMSR), change from baseline of JAK2 mutated allele burden.
Response Assessment in Study Participants With ET | Up to 1 year in Phase 1c
  Response will be evaluated according to ELN and 2013 IWG-MRT criteria, including ORR, DOR, TTR, PFS, percentage of study participants who achieved CHR, duration of CHR, percentage of study participants with >50% change in MPN-SAF TSS, percentage of study participants who achieve SVR35 from baseline, DoMSR, change from baseline of JAK2 mutated allele burden.
Response Assessment in Study Participants With MF | Up to 1 year in Phase 1c
  Response will be evaluated according to the European Myelofibrosis Network (EUMNET) and 2013 IWG-MRT criteria, including ORR, DOR, TTR, PFS, percentage of study participants who achieve anemia response, percentage of study participants with symptom response, percentage of study participants who achieve SVR35 from baseline, DoMSR, change from baseline of JAK2 mutated allele burden.
Response Assessment in Study Participants With LR-MDS | Up to 1 year in Phase 1c
  Response will be evaluated according to the 2006 Myelodysplastic Syndromes International Council for Harmonisation (MDS-IWG) criteria, including percentage of study participants with hematology improvement (HI) (erythroid/platelet/neutrophil responses), percentage of study participants with complete response (CR), partial response (PR) or marrow complete response (mCR), DOR, TTR, PFS, percentage of study participants who achieve red blood cell transfusion independence (RBC-TI) ≥ 8 weeks, time to RBC-TI and duration of RBC-TI for study participants who achieve RBC TI ≥ 8 weeks on treatment.
Response Assessment in Study Participants With HR-MDS | Up to 1 year in Phase 1c
  Response was evaluated according to the 2006 MDS-IWG criteria, including HI (erythroid/platelet/neutrophil responses), percentage of study participants with CR, PR or mCR, DOR, TTR, PFS, minimal residual disease (MRD) monitoring in participants who achieve CR.
Response Assessment in Study Participants With AML | Up to 1 year in Phase 1c
  Response was evaluated according to the 2022 ELN for AML criteria, including CR, CR with incomplete hematologic recovery (CRi), CR with partial hematological recovery (CRh), morphologic leukemia-free state (MLFS), percentage of study participants with PR, DOR, TTR, event-free survival (EFS), MRD monitoring in study participants who achieve CR/CRi/CRh.

SECONDARY OUTCOMES:
GLB-001 and GLB-C183-A-2 (diastereoisomer of GLB-001) Pharmacokinetics after Single Administration - AUC0-last | Up to 48 hours after single administration
  Area under the concentration-time curve from zero to the last measurable concentration.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Single Administration - AUC0-24 | Up to 48 hours after single administration
  Area under the concentration-time curve from 0 to 24 hours.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Single Administration - AUC0-inf | Up to 48 hours after single administration
  Area under the concentration-time curve from 0 to infinity.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Single Administration - Cmax | Up to 48 hours after single administration
  Maximum plasma concentration.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Single Administration - Tmax | Up to 48 hours after single administration
  The time to reach maximum concentration.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Single Administration - T1/2 | Up to 48 hours after single administration
  Terminal half-life.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Single Administration - Vz/F | Up to 48 hours after single administration
  Apparent volume of distribution.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Single Administration - CL/F | Up to 48 hours after single administration
  Apparent total clearance of the drug from plasma after oral administration.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Single Administration - λz | Up to 48 hours after single administration
  Terminal rate constant.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Multiple Administration - Tmax,ss | Up to 1 year
  Time of maximum concentration at steady state.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Multiple Administration - Cav,ss | Up to 1 year
  Average plasma concentration at steady state.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Multiple Administration - Cmax,ss | Up to 1 year
  Maximum plasma concentration at steady state.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Multiple Administration - Cmin,ss | Up to 1 year
  Minimum plasma concentration at steady state.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Multiple Administration - AUC0-tau | Up to 1 year
  Area under the concentration-time curve during the dosing interval.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Multiple Administration-AUC0-last | Up to 1 year
  Area under the concentration-time curve from zero to the last measurable concentration.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Multiple Administration - λz | Up to 1 year
  Terminal rate constant.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Multiple Administration - Vz/F | Up to 1 year
  Apparent volume of distribution.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Multiple Administration - CLss/F | Up to 1 year
  Apparent clearance at steady state.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Multiple Administration - T1/2 | Up to 1 year
  Terminal half-life.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Multiple Administration - Rac [AUC] | Up to 1 year
  Accumulation index in area under the concentration-time curve.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Multiple Administration - Rac [Cmax] | Up to 1 year
  Accumulation index in maximum plasma concentration.
GLB-001 and GLB-C183-A-2 Pharmacokinetics after Multiple Administration-DF | Up to 1 year
  Degree of fluctuation index.

CONTACTS AND LOCATIONS:
Overall Officials: Gang Lu, Ph.D., Study Director — Hangzhou GluBio Pharmaceutical Co., Ltd.
Locations (14):
- China (14):
  - The First Affiliated Hospital of University of Science and Technology of China (Anhui Provincial Hospital), Hefei, Anhui
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality
  - The First Hospital of Hebei Medical Universtiy, Shijiazhuang, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Zhongnan Hospital of Wuhan University, Wuhan, Hubei
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - Sheng Jing Hospital of China Medical Universtiy, Shenyang, Liaoning
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Institute of Hematology and Blood Diseases Hospital, Chinese Academy of Medical Sciences, Tianjin, Tianjin Municipality
  - The Second Hospital of Tianjin Medical Universtiy, Tianjin, Tianjin Municipality
  - The First Affilicated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - The First Affiliated Hospital of Wenzhou Medical University, Wenzhou, Zhejiang